CLINICAL TRIAL: NCT04958733
Title: Does Bone Grafting at the Time of Bone-Patellar Tendon-Bone ACL Reconstruction Reduce the Incidence of Post-operative Anterior Knee Pain: A Randomized Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHC-2021-0113
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Bone Grafting (Active Comparator): Excess bone obtained from graft preparation and the coring reamer will be used to fill the patellar and tibial donor sites.
  Interventions: Procedure: Autologous bone grafting
- Control (Placebo Comparator): The control group will have their patellar and tibial defects remain unfilled.
  Interventions: Procedure: Absence of autologous bone grafting

INTERVENTIONS:
Procedure: Autologous bone grafting — Autologous bone grafting is the excess bone obtained from graft preparation and the coring reamer
  Arms: Autologous Bone Grafting
Procedure: Absence of autologous bone grafting — Donor sites will be left unfilled
  Arms: Control

SUMMARY:
It is estimated that 48 out of 10,000 people, in the United States, will tear their anterior cruciate ligament (ACL) annually and undergo ACL reconstruction (ACLR). Surgeons have several graft options, surgical techniques, and fixation methods to consider when planning how to reconstruct a patient's ACL. Graft options vary greatly and include allografts and autografts with good evidence that are good choices. Further, autografts include several different specific grafts including; bone-patellar tendon-bone (BPTB), hamstring tendons, and quadriceps tendon. There is no clear consensus on which graft type is superior, as each graft has associated positives and negatives.

Historically, autologous BPTB grafts have been the preferred choice of surgeons given its ability to restore rotational stability for the knee, the robust healing with direct bone-to-bone contact at both ends of the graft, and low failure rates. However, there are drawbacks to ACLR using a BPTB graft. Complications following BPTB graft harvesting include patella fractures, patellar tendon ruptures, increased risk of patellofemoral osteoarthritis, lack of terminal extension, and donor-site morbidity. The majority of these complications are associated with low-risk rates, except for donor-site morbidity which may be prevalent in 37-51% of BPTB graft patients. Donor-site pain can manifest as anterior knee, patellofemoral pain, loss of sensory input, or discomfort with kneeling and can negatively influence subjective as well as objective measures of knee function.

Filling bony defects with bone graft is a procedure that is commonly conducted within orthopedics. However, its use in treating the bony defects caused during BPTB graft harvesting is less common as patella and tibial harvest sites are routinely left unfilled. Significant methodological differences in treatment interventions for the patella harvest site, the tibial harvest site, or both and conflicting results have made it difficult to determine if these treatments have clinical utility. To the best of the investigators' knowledge, there has been no investigation looking at the incidence of donor site morbidity treated with autologous bone grafting of the harvest sites. Therefore, the purpose of this study is to determine if filling the harvest site defect is associated with a lower rate of donor site morbidity and better patient reported functional outcomes compared to patients whose harvest site remains unfilled.

The purpose of this study is to compare the rate of donor site morbidity between patients who have their harvest sites bone grafted with autologous bone (BG) and those whose harvest sites remain unfilled (nBG).

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18 years of age and older, with no upper age limit
* A candidate for primary autologous BPTB ACLR
* Willing to participate in the study

Exclusion Criteria:

* Concomitant ligamentous or chondral injury
* Prior surgery on the index knee
* Prior history of anterior knee pain or patellofemoral joint pain on the index knee
* Outerbridge classification > 2 assessed during arthroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | pre-op
  The Visual Analog Scale (VAS) is a 10-cm line that allows subjects to visually report their pain between "no pain" (0 cm) on the left and "constant pain" (10 cm) on the right. Patients will be asked to complete the VAS with the prompt, "Please indicate the amount of pain you are feeling right now in the front of your knee." It is considered a worse outcome the closer the patient marks to the "constant pain" on the right of the scale.
Visual Analog Scale | post-op month 6
  The Visual Analog Scale (VAS) is a 10-cm line that allows subjects to visually report their pain between "no pain" (0 cm) on the left and "constant pain" (10 cm) on the right. Patients will be asked to complete the VAS with the prompt, "Please indicate the amount of pain you are feeling right now in the front of your knee." It is considered a worse outcome the closer the patient marks to the "constant pain" on the right of the scale.
Visual Analog Scale | post-op month 12
  The Visual Analog Scale (VAS) is a 10-cm line that allows subjects to visually report their pain between "no pain" (0 cm) on the left and "constant pain" (10 cm) on the right. Patients will be asked to complete the VAS with the prompt, "Please indicate the amount of pain you are feeling right now in the front of your knee." It is considered a worse outcome the closer the patient marks to the "constant pain" on the right of the scale.
Visual Analog Scale | post-op month 24
  The Visual Analog Scale (VAS) is a 10-cm line that allows subjects to visually report their pain between "no pain" (0 cm) on the left and "constant pain" (10 cm) on the right. Patients will be asked to complete the VAS with the prompt, "Please indicate the amount of pain you are feeling right now in the front of your knee." It is considered a worse outcome the closer the patient marks to the "constant pain" on the right of the scale.
Direct Palpation of Harvest Site | pre-op
  Subjects will be asked to rate their pain as either 'no pain', 'mild pain' or 'sharp pain' during direct palpation for both the patella and tibial harvest sites. 'Sharp pain' is considered the worse outcome, 'mild pain' as a median outcome, and 'no pain' is considered the best outcome of the three.
Direct Palpation of Harvest Site | post-op month 6
  Subjects will be asked to rate their pain as either 'no pain', 'mild pain' or 'sharp pain' during direct palpation for both the patella and tibial harvest sites. 'Sharp pain' is considered the worse outcome, 'mild pain' as a median outcome, and 'no pain' is considered the best outcome of the three.
Direct Palpation of Harvest Site | post-op month 12
  Subjects will be asked to rate their pain as either 'no pain', 'mild pain' or 'sharp pain' during direct palpation for both the patella and tibial harvest sites. 'Sharp pain' is considered the worse outcome, 'mild pain' as a median outcome, and 'no pain' is considered the best outcome of the three.
Direct Palpation of Harvest Site | post-op month 24
  Subjects will be asked to rate their pain as either 'no pain', 'mild pain' or 'sharp pain' during direct palpation for both the patella and tibial harvest sites. 'Sharp pain' is considered the worse outcome, 'mild pain' as a median outcome, and 'no pain' is considered the best outcome of the three.
Pain with Kneeling | pre-op
  Subjects will also be asked to kneel on the floor of the examination room and rate their pain as either 'no pain', 'mild pain', 'unable to kneel on hard surface but able with cushion/pad', or 'complete inability to kneel'. 'Complete inability to kneel' is considered the worst outcome within this measure, with the following considered increasing better outcomes in this order: 'unable to kneel on hard surface but able with cushion/pad', 'mild pain', 'no pain'.
Pain with Kneeling | post-op month 6
  Subjects will also be asked to kneel on the floor of the examination room and rate their pain as either 'no pain', 'mild pain', 'unable to kneel on hard surface but able with cushion/pad', or 'complete inability to kneel'. 'Complete inability to kneel' is considered the worst outcome within this measure, with the following considered increasing better outcomes in this order: 'unable to kneel on hard surface but able with cushion/pad', 'mild pain', 'no pain'.
Pain with Kneeling | post-op month 12
  Subjects will also be asked to kneel on the floor of the examination room and rate their pain as either 'no pain', 'mild pain', 'unable to kneel on hard surface but able with cushion/pad', or 'complete inability to kneel'. 'Complete inability to kneel' is considered the worst outcome within this measure, with the following considered increasing better outcomes in this order: 'unable to kneel on hard surface but able with cushion/pad', 'mild pain', 'no pain'.
Pain with Kneeling | post-op month 24
  Subjects will also be asked to kneel on the floor of the examination room and rate their pain as either 'no pain', 'mild pain', 'unable to kneel on hard surface but able with cushion/pad', or 'complete inability to kneel'. 'Complete inability to kneel' is considered the worst outcome within this measure, with the following considered increasing better outcomes in this order: 'unable to kneel on hard surface but able with cushion/pad', 'mild pain', 'no pain'.

SECONDARY OUTCOMES:
PROMIS-10 | pre-op
  The Patient-Reported Outcomes Measurement Information System-10 (PROMIS-10) will be used to assess global quality of health. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
PROMIS-10 | post-op month 6
  The Patient-Reported Outcomes Measurement Information System-10 (PROMIS-10) will be used to assess global quality of health. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
PROMIS-10 | post-op month 12
  The Patient-Reported Outcomes Measurement Information System-10 (PROMIS-10) will be used to assess global quality of health. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
PROMIS-10 | post-op month 24
  The Patient-Reported Outcomes Measurement Information System-10 (PROMIS-10) will be used to assess global quality of health. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
International Knee Documentation Committee (IKDC) Subjective form | pre-op
  The International Knee Documentation Committee (IKCD) subjective form will be used to assess knee-specific functional abilities. The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
International Knee Documentation Committee (IKDC) Subjective form | post-op month 6
  The International Knee Documentation Committee (IKCD) subjective form will be used to assess knee-specific functional abilities. The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
International Knee Documentation Committee (IKDC) Subjective form | post-op month 12
  The International Knee Documentation Committee (IKCD) subjective form will be used to assess knee-specific functional abilities. The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
International Knee Documentation Committee (IKDC) Subjective form | post-op 24
  The International Knee Documentation Committee (IKCD) subjective form will be used to assess knee-specific functional abilities. The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) | pre-op
  The Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) will be used to assess functional limitations due to patellofemoral joint pain. This will be necessary to evaluate as the BPBT graft is harvested from the patellar and may affect the function of the patellofemoral joint. KOOS-PF is an 11 item patient reported outcome, with each item rated as Never/none = 0, Monthly/mild = 1, Weekly/moderate = 2, Daily/severe = 3, Always/extreme = 4. The mean score is calculated for the 11 items, and divided by the maximum possible score for each item (i.e. 4). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.
Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) | post-op month 6
  The Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) will be used to assess functional limitations due to patellofemoral joint pain. This will be necessary to evaluate as the BPBT graft is harvested from the patellar and may affect the function of the patellofemoral joint. KOOS-PF is an 11 item patient reported outcome, with each item rated as Never/none = 0, Monthly/mild = 1, Weekly/moderate = 2, Daily/severe = 3, Always/extreme = 4. The mean score is calculated for the 11 items, and divided by the maximum possible score for each item (i.e. 4). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.
Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) | post-op month 12
  The Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) will be used to assess functional limitations due to patellofemoral joint pain. This will be necessary to evaluate as the BPBT graft is harvested from the patellar and may affect the function of the patellofemoral joint. KOOS-PF is an 11 item patient reported outcome, with each item rated as Never/none = 0, Monthly/mild = 1, Weekly/moderate = 2, Daily/severe = 3, Always/extreme = 4. The mean score is calculated for the 11 items, and divided by the maximum possible score for each item (i.e. 4). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.
Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) | post-op month 24
  The Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF) will be used to assess functional limitations due to patellofemoral joint pain. This will be necessary to evaluate as the BPBT graft is harvested from the patellar and may affect the function of the patellofemoral joint. KOOS-PF is an 11 item patient reported outcome, with each item rated as Never/none = 0, Monthly/mild = 1, Weekly/moderate = 2, Daily/severe = 3, Always/extreme = 4. The mean score is calculated for the 11 items, and divided by the maximum possible score for each item (i.e. 4). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.
Marx Activity Scale | pre-op
  The Marx Activity scale will be used to assess frequency and intensity of athletic participation. The Marx Scale consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year. The maximum score is 16 points, the closer the score is to 16 the higher the intensity and frequency of activity.
Marx Activity Scale | post-op month 6
  The Marx Activity scale will be used to assess frequency and intensity of athletic participation. The Marx Scale consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year. The maximum score is 16 points, the closer the score is to 16 the higher the intensity and frequency of activity.
Marx Activity Scale | post-op month 12
  The Marx Activity scale will be used to assess frequency and intensity of athletic participation. The Marx Scale consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year. The maximum score is 16 points, the closer the score is to 16 the higher the intensity and frequency of activity.
Marx Activity Scale | post-op month 24
  The Marx Activity scale will be used to assess frequency and intensity of athletic participation. The Marx Scale consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year. The maximum score is 16 points, the closer the score is to 16 the higher the intensity and frequency of activity.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bone and Joint Institute at Hartford Hospital, Hartford, Connecticut
  - Orthopedic Associates of Hartford, Hartford, Connecticut
  - PRISM Sports Medicine, Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers at this time.

REFERENCES:
- [Result] Ahn JH, Kim JG, Wang JH, Jung CH, Lim HC. Long-term results of anterior cruciate ligament reconstruction using bone-patellar tendon-bone: an analysis of the factors affecting the development of osteoarthritis. Arthroscopy. 2012 Aug;28(8):1114-23. doi: 10.1016/j.arthro.2011.12.019. Epub 2012 Mar 13. PMID 22421565
- [Result] Brown K, Solomon MJ, Young J, Seco M, Bannon PG. Addressing the ethical grey zone in surgery: a framework for identification and safe introduction of novel surgical techniques and procedures. ANZ J Surg. 2019 Jun;89(6):634-638. doi: 10.1111/ans.15104. Epub 2019 Apr 11. PMID 30974516
- [Result] Brydone AS, Meek D, Maclaine S. Bone grafting, orthopaedic biomaterials, and the clinical need for bone engineering. Proc Inst Mech Eng H. 2010 Dec;224(12):1329-43. doi: 10.1243/09544119JEIM770. PMID 21287823
- [Result] Cervellin M, de Girolamo L, Bait C, Denti M, Volpi P. Autologous platelet-rich plasma gel to reduce donor-site morbidity after patellar tendon graft harvesting for anterior cruciate ligament reconstruction: a randomized, controlled clinical study. Knee Surg Sports Traumatol Arthrosc. 2012 Jan;20(1):114-20. doi: 10.1007/s00167-011-1570-5. Epub 2011 Jun 16. PMID 21678095
- [Result] Kartus J, Stener S, Lindahl S, Engstrom B, Eriksson BI, Karlsson J. Factors affecting donor-site morbidity after anterior cruciate ligament reconstruction using bone-patellar tendon-bone autografts. Knee Surg Sports Traumatol Arthrosc. 1997;5(4):222-8. doi: 10.1007/s001670050054. PMID 9430571
- [Result] Leathers MP, Merz A, Wong J, Scott T, Wang JC, Hame SL. Trends and Demographics in Anterior Cruciate Ligament Reconstruction in the United States. J Knee Surg. 2015 Oct;28(5):390-4. doi: 10.1055/s-0035-1544193. Epub 2015 Jan 30. PMID 25635874
- [Result] Mastrokalos DS, Springer J, Siebold R, Paessler HH. Donor site morbidity and return to the preinjury activity level after anterior cruciate ligament reconstruction using ipsilateral and contralateral patellar tendon autograft: a retrospective, nonrandomized study. Am J Sports Med. 2005 Jan;33(1):85-93. doi: 10.1177/0363546504265926. PMID 15611003
- [Result] Schandl K, Horvathy DB, Doros A, Majzik E, Schwarz CM, Csonge L, Abkarovits G, Bucsi L, Lacza Z. Bone-Albumin filling decreases donor site morbidity and enhances bone formation after anterior cruciate ligament reconstruction with bone-patellar tendon-bone autografts. Int Orthop. 2016 Oct;40(10):2097-2104. doi: 10.1007/s00264-016-3246-8. Epub 2016 Jun 29. PMID 27357530
- [Result] Walters BL, Porter DA, Hobart SJ, Bedford BB, Hogan DE, McHugh MM, Klein DA, Harousseau K, Nicholas SJ. Effect of Intraoperative Platelet-Rich Plasma Treatment on Postoperative Donor Site Knee Pain in Patellar Tendon Autograft Anterior Cruciate Ligament Reconstruction: A Double-Blind Randomized Controlled Trial. Am J Sports Med. 2018 Jul;46(8):1827-1835. doi: 10.1177/0363546518769295. Epub 2018 May 9. PMID 29741923
- [Result] Xie X, Liu X, Chen Z, Yu Y, Peng S, Li Q. A meta-analysis of bone-patellar tendon-bone autograft versus four-strand hamstring tendon autograft for anterior cruciate ligament reconstruction. Knee. 2015 Mar;22(2):100-10. doi: 10.1016/j.knee.2014.11.014. Epub 2014 Dec 11. PMID 25547048